CLINICAL TRIAL: NCT04760314
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Lebrikizumab When Used in Combination With Topical Corticosteroid Treatment in Japanese Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study of Lebrikizumab (LY3650150) in Combination With Topical Corticosteroids in Japanese Participants With Moderate-to-Severe Atopic Dermatitis
Acronym: ADhere-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17953; J2T-JE-KGAL (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Skin Diseases, Genetic
Keywords: Corticosteroids
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Skin Diseases, Genetic | interventions — lebrikizumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lebrikizumab 250 mg Every 4 weeks (Q4W) (Experimental): Participants received 500 mg of Lebrikizumab (2 x 250 mg) subcutaneous (SC) injections as a loading dose at Baseline followed by 250 mg of Lebrikizumab administered SC Q4W from Week 4 until Week 12, in combination with topical corticosteroid. Week 16 responders entered maintenance period and continued with the same treatment. Week 16 non responders entered Escape Arm and received Lebrikizumab 250 mg Q2W until Week 68.
  Interventions: Drug: Lebrikizumab; Drug: Topical Corticosteroid
- Lebrikizumab 250 mg Every 2 weeks (Q2W) (Experimental): Participants received 500 mg of Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 followed by 250 mg of Lebrikizumab administered SC Q2W from Week 4 until Week 14, in combination with topical corticosteroid. Week 16 responders entered maintenance period and were randomly allocated to receive 250 mg lebrikizumab Q2W or 250 mg lebrikizumab Q4W, in a 1:1 ratio. Week 16 non responders entered Escape Arm and received Lebrikizumab 250 mg Q2W until Week 68.
  Interventions: Drug: Lebrikizumab; Drug: Topical Corticosteroid
- Placebo (Placebo Comparator): Participants received two SC injections of Placebo as a loading dose at Baseline in combination with topical corticosteroid and Week 2 followed by a single injection Q2W from Week 4 until Week 14. Week 16 responders entered maintenance period and continued with the same treatment. Week 16 non responders entered Escape Arm and received Lebrikizumab 250 mg Q2W until Week 68.
  Interventions: Drug: Placebo; Drug: Topical Corticosteroid

INTERVENTIONS:
Drug: Lebrikizumab — Administered SC
  Other Names: LY3650150
  Arms: Lebrikizumab 250 mg Every 2 weeks (Q2W); Lebrikizumab 250 mg Every 4 weeks (Q4W)
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Topical Corticosteroid — Self-applied

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of lebrikizumab in combination with a topical corticosteroids in Japanese participants with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic Atopic Dermatitis (AD) that has been present for ≥1 year before the screening.
* Have moderate-to-severe AD, including all of the following:

  * EASI score ≥16 at the baseline
  * IGA score ≥3 (scale of 0 to 4) at the baseline
  * AD involvement on ≥10% of Body Surface Area (BSA) at the baseline
* Have a documented history provided by a physician and/or investigator of inadequate response to existing topical medications within 6 months preceding screening as defined by at least 1 of the following:

  * Inability to achieve good disease control, defined as mild disease or better (for example, IGA ≤2) after use of at least a medium-potency topical corticosteroids (TCS) for at least 4 weeks, or for the maximum duration recommended by the product prescribing information (for example, 14 days for super-potent TCS), whichever is shorter. Topical corticosteroids may be used with or without Topical calcineurin inhibitors (TCI) and/or topical Janus Kinase (JAK) inhibitors.
  * Participants who failed systemic therapies intended to treat AD within 6 months preceding screening, such as cyclosporine, methotrexate (MTX), azathioprine, and mycophenolate mofetil (MMF), will also be considered as surrogates for having inadequate response to topical therapy.
* Body weight ≥40 kilogram (kg)

Exclusion Criteria:

* Have a history of anaphylaxis
* Have uncontrolled chronic disease that might require bursts of oral corticosteroids for example, comorbid severe uncontrolled asthma within the past 12 months requiring systemic corticosteroid treatment or hospitalization for >24 hours at baseline.
* Have an active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline or superficial skin infections within 1 week before the baseline.
* Evidence of acute or chronic hepatitis or known liver cirrhosis.
* Have a history of pneumocystis pneumonia (PCP) or a positive beta-D-glucan test at screening and a confirmed diagnosis of PCP.
* Have a history of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* Have presence of skin comorbidities (for example, sclerosis, psoriasis, or lupus erythematosus) that may interfere with study assessments.
* Have presence of significant uncontrolled neuropsychiatric disorder.
* Have been exposed to a live vaccine within 12 weeks prior to baseline or are expected to need/receive a live vaccine during the study or up to 125 days after the last dose of study drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- Japan (37):
  - Yanagihara dermatology clinic, Ainokawa, Ichikawa-shi, Chiba
  - Kawashima Dermatology Clinic, Ichikawa-shi, Chiba
  - Charme Clinique, Matsudo, Chiba
  - Yasumoto Dermatology Clinic, Chikushino-shi, Fukuoka
  - Hino Dermatology Clinic, Fukutsu, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Takagi Dermatology, Obihiro, Hokkaido
  - Sapporo Skin Clinic, Sapporo, Hokkaido
  - Kobayashi Skin Clinic, Sapporo, Hokkaido
  - Dermatology Shimizu Clinic, Kobe, Hyōgo
  - Ibaraki Medical Center, Inashiki-gun, Ibaraki
  - KAJI Dermatology Clinic, Nonoichi-shi, Ishikawa-ken
  - Kosugi Dermatology Clinic, Kawasaki, Kanagawa
  - Queen's Square Dermatology and Allergology, Nishi-ku, Yokohama-city, Kanagawa
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Noguchi Dermatology, Kashima-machi, Kamimashiki-gun, Kumamoto
  - Jyouzanhihuka・Hinyoukika Clinic, Kumamoto, Kumamoto
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Mochida Dermatology Clinic, Izumiotsu-shi, Osaka
  - Kume Clinic, Sakai, Osaka
  - Yoshikawa Dermatology Clinic, Takatsuki, Osaka
  - Sanrui Dermatology Clinic, Ohmiya-ku,Saitama-shi, Saitama
  - Dokkyo Medical University Hospital, Shimotsuga-Gun, Tochigi
  - Akihabara Skin Clinic, Chiyoda-ku, Tokyo
  - Sumire Dermatology Clinic, Edogawa-ku, Tokyo
  - Maruyama Dermatology Clinic, Koto-ku, Tokyo
  - Hamaguchi Skin Clinic, Machida-shi, Tokyo
  - Mita Dermatology Clinic, Minato-Ku, Tokyo
  - Tanpopo Dermatology Clinic, Ōta-ku, Tokyo
  - Yamate Dermatological Clinic, Shinjuku, Tokyo
  - Yoshihara Dermatology Clinic, Sumida-ku, Tokyo
  - Tachikawa Dermatology Clinic, Tachikawa-shi, Tokyo
  - Shirasaki Clinic, Takaoka-shi, Toyama
  - Matsuda Tomoko Dermatological Clinic, Fukuoka
  - Kyoto Furitsu Medical University Hospital, Kyoto
  - Osaka City University Hospital, Osaka
  - Goto Dermatology Clinic, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Katoh N, Tanaka A, Takahashi H, Shimizu R, Kataoka Y, Torisu-Itakura H, Morisaki Y, Yamamoto C, Igawa K. Long-term management of moderate-to-severe atopic dermatitis with lebrikizumab and concomitant topical corticosteroids: a 68-week randomized double-blind placebo-controlled phase III trial in Japan (ADhere-J). Br J Dermatol. 2025 Mar 18;192(4):597-610. doi: 10.1093/bjd/ljae394. PMID 39442013
- See also: A Study of Lebrikizumab (LY3650150) in Combination With Topical Corticosteroids in Japanese Participants With Moderate-to-Severe Atopic Dermatitis (ADhere-J) — https://trials.lillytrialguide.com/en-US/trial/6Snw910hnAdavPQabysPCL

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Induction period (16-weeks): Participants were randomly assigned to 250mg Lebrikizumab every 2 weeks (Q2W) or 250mg Lebrikizumab every 4 weeks (Q4W) or Placebo.
  Maintenance period (52-weeks): At week 16, responders from 250mg Lebrikizumab Q2W were re-randomised to 250mg Lebrikizumab Q2W and 250mg Lebrikizumab Q4W; responders from 250mg Lebrikizumab Q4W or Placebo arms continued with same treatment. Responders were defined as having an IGA of 0 or 1 or a 75% reduction in EASI (EASI-75).
Pre-assignment Details: (continued) Escape arm: Induction non-responder (i.e.) participants who do not achieve an IGA of 0 or 1 or an EASI-75 at Week 16 and maintenance non-responders (i.e.) those not maintaining an EASI-50 response at week 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, or 64 following week 16 were assigned to an Escape Arm and received lebrikizumab 250 mg as open-label treatment Q2W through Week 68.
  Throughout the trial, participants received the study drug in combination with topical corticosteroid.
Groups:
- Induction - Placebo: Induction Period: (Baseline - Week 16): Participants received two subcutaneous (SC) injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection Q2W from Week 4 until Week 14.
- Induction - Lebrikizumab 250mg Q4W: Induction Period (Baseline - Week 16): Participants received 500 mg of Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline followed by 250 mg of Lebrikizumab administered SC Q4W from Week 4 until Week 12.
- Induction - Lebrikizumab 250mg Q2W: Induction Period (Baseline - Week 16): Participants received 500 mg of Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 followed by 250 mg of Lebrikizumab administered SC Q2W from Week 4 until Week 14.
- Maintenance Blinded Period - Placebo Responder/Placebo: Maintenance Secondary Population:
  Maintenance Period (Week 16 - Week 68): Participants received Placebo administered SC Q2W from Week 16 to Week 66.
- Maintenance Blinded Period - Lebrikizumab Q4W Responder/Lebrikizumab Q4W: Maintenance Primary Population:
  Maintenance Period (Week 16 - Week 68): Participants received 250 mg Lebrikizumab administered SC Q4W from Weeks 16 until Week 64.
- Maintenance Blinded Period - Lebrikizumab Q2W Responder/ Lebrikizumab Q4W: Maintenance Primary Population:
  Maintenance Period (Week 16 - Week 68): Participants received 250 mg Lebrikizumab administered SC Q4W from Week 16 until Week 64.
- Maintenance Blinded Period - Lebrikizumab Q2W Responder/Lebrikizumab Q2W: Maintenance Period (Week 16 - Week 68): Participants received 250 mg of Lebrikizumab administered SC Q2W from Week 16 until Week 66.
- Escape Arm Week 16 - Maintenance Open Label - Placebo Non Responder/Lebrikizumab 250 mg Q2W: Participants received blinded doses based on prior treatment assignment followed by one 250 mg Lebrikizumab administered SC Q2W until Week 68 in an open-label fashion.
  For participants who received placebo in the Induction Period, loading dose was:
  Two 250 mg Lebrikizumab SC injection on Week 16 and two 250 mg Lebrikizumab SC injections on Week 18.
  For participants who did not maintain an acceptable response during the Maintenance Period and entered the Escape Arm, the loading doses were administrated at entry and 2 weeks after entry based on the treatment assignment prior to entering escape arm.
- Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q4W Nonresponder/Lebrikizumab 250mg Q2W: Participants received blinded doses based on prior treatment assignment followed by one 250 mg Lebrikizumab administered SC Q2W until Week 68 in an open-label fashion.
  For participants who received Lebrikizumab Q4W in the Induction Period, the loading dose was:
  One 250 mg Lebrikizumab administered SC on Week16 and Week 18. For participants who did not maintain an acceptable response during the Maintenance Period and entered the Escape Arm, the loading doses were administrated at entry and 2 weeks after entry based on the treatment assignment prior to entering escape arm.
- Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q2W Nonresponder/Lebrikizumab 250mg Q2W: Participants received blinded doses based on prior treatment assignment followed by one 250 mg Lebrikizumab administered SC Q2W until Week 68 in an open-label fashion.
  For participants who received Lebrikizumab Q2W in the Induction Period, the loading dose was:
  One 250 mg Lebrikizumab administered SC on Week16 and Week 18. For participants who did not maintain an acceptable response during the Maintenance Period and entered the Escape Arm, the loading doses were administrated at entry and 2 weeks after entry based on the treatment assignment prior to entering escape arm.
- Escape Arm Week 20 to 64 Maintenance Open Label Lebrikizumab 250 Q2W: Participants received 250 mg Lebrikizumab administered SC Q2W through Week 68 in an open-label fashion.
Period: Induction Period
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250mg Q4W | Induction - Lebrikizumab 250mg Q2W | Maintenance Blinded Period - Placebo Responder/Placebo | Maintenance Blinded Period - Lebrikizumab Q4W Responder/Lebrikizumab Q4W | Maintenance Blinded Period - Lebrikizumab Q2W Responder/ Lebrikizumab Q4W | Maintenance Blinded Period - Lebrikizumab Q2W Responder/Lebrikizumab Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Non Responder/Lebrikizumab 250 mg Q2W | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q4W Nonresponder/Lebrikizumab 250mg Q2W | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q2W Nonresponder/Lebrikizumab 250mg Q2W | Escape Arm Week 20 to 64 Maintenance Open Label Lebrikizumab 250 Q2W
Started | 82 | 81 | 123 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 82 | 81 | 123 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 82 (Completed includes Responders n = 11; Non responders n = 71.) | 80 (Completed includes Responders n = 38; Non responders n = 42.) | 120 (Completed includes Responders n = 65; Non responders n = 55.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Blinded Period
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250mg Q4W | Induction - Lebrikizumab 250mg Q2W | Maintenance Blinded Period - Placebo Responder/Placebo | Maintenance Blinded Period - Lebrikizumab Q4W Responder/Lebrikizumab Q4W | Maintenance Blinded Period - Lebrikizumab Q2W Responder/ Lebrikizumab Q4W | Maintenance Blinded Period - Lebrikizumab Q2W Responder/Lebrikizumab Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Non Responder/Lebrikizumab 250 mg Q2W | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q4W Nonresponder/Lebrikizumab 250mg Q2W | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q2W Nonresponder/Lebrikizumab 250mg Q2W | Escape Arm Week 20 to 64 Maintenance Open Label Lebrikizumab 250 Q2W
Started | 0 (Participants were assigned to this arm only during Induction Period.) | 0 (Participants were assigned to this arm only during Induction Period.) | 0 (Participants were assigned to this arm only during Induction Period.) | 11 (Only those participants who responded to Induction Placebo or Lebrikizumab at Week 16 entered the Maintenance Period.) | 38 (Only those participants who responded to Induction Placebo or Lebrikizumab at Week 16 entered the Maintenance Period.) | 33 (Only those participants who responded to Induction Placebo or Lebrikizumab at Week 16 entered the Maintenance Period.) | 32 (Only those participants who responded to Induction Placebo or Lebrikizumab at Week 16 entered the Maintenance Period.) | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 11 | 38 | 33 | 32 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 9 | 35 | 27 | 27 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 3 | 6 | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Enrolled to Escape Arm | 0 | 0 | 0 | 1 | 0 | 4 | 3 | 0 | 0 | 0 | 0
Not completed — Assigned Treatment by Mistake | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Open Label Escape Arm
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250mg Q4W | Induction - Lebrikizumab 250mg Q2W | Maintenance Blinded Period - Placebo Responder/Placebo | Maintenance Blinded Period - Lebrikizumab Q4W Responder/Lebrikizumab Q4W | Maintenance Blinded Period - Lebrikizumab Q2W Responder/ Lebrikizumab Q4W | Maintenance Blinded Period - Lebrikizumab Q2W Responder/Lebrikizumab Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Non Responder/Lebrikizumab 250 mg Q2W | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q4W Nonresponder/Lebrikizumab 250mg Q2W | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q2W Nonresponder/Lebrikizumab 250mg Q2W | Escape Arm Week 20 to 64 Maintenance Open Label Lebrikizumab 250 Q2W
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 71 (Only those participants who did not respond to Induction Placebo or Lebrikizumab entered Escape Arm at Week 16.) | 42 (Only those participants who did not respond to Induction Placebo or Lebrikizumab entered Escape Arm at Week 16.) | 55 (Only those participants who did not respond to Induction Placebo or Lebrikizumab entered Escape Arm at Week 16.) | 8 (Only those participants who did not respond to treatment during maintenance period (i.e.) not maintaining an EASI-50 response at Weeks 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, or 64 were entered here.)
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 71 | 42 | 55 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63 | 40 | 48 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 7 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 5 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Induction - Placebo: Induction Period: (Baseline - Week 16): Participants received two SC injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection Q2W from Week 4 until Week 14.
- Induction - Lebrikizumab 250 mg Q4W: Induction Period (Baseline - Week 16): Participants received 500 mg of Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline followed by 250 mg of Lebrikizumab administered SC Q4W from Week 4 until Week 12.
- Induction - Lebrikizumab 250 mg Q2W: Induction Period (Baseline - Week 16): Participants received 500 mg of Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 followed by 250 mg of Lebrikizumab administered SC Q2W from Week 4 until Week 14.
- Total: Total of all reporting groups
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W | Total
Number analyzed (Participants) | 82 | 81 | 123 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.80 (13.60) | 37.80 (12.02) | 35.50 (12.24) | 36.00 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 41 | 90
  Male | 58 | 56 | 82 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 82 | 81 | 123 | 286
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 82 | 81 | 123 | 286
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 82 | 81 | 123 | 286

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Investigators Global Assessment (IGA) Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 16
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Baseline to Week 16
Population: All randomized participants, even if the participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Markov Chain Monte Carlo Multiple Imputation (MCMC-MI) was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 82 | 81 | 123
Percentage of participants | 6.1 [0.9 to 11.3] | 29.1 [19.2 to 39.1] | 33.4 [25.0 to 41.8]
Statistical Analysis 1: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 22.6, 95% CI 2-sided [11.6 to 33.6]
Statistical Analysis 2: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q2W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 27.3, 95% CI 2-sided [17.5 to 37.0]

2. Primary Outcome: Percentage of Participants Achieving Eczema Area Severity Index-75 (EASI-75) (≥75% Reduction in EASI Score) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI-75 score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 82 | 81 | 123
Percentage of participants | 13.4 [6.0 to 20.8] | 47.2 [36.3 to 58.1] | 51.2 [42.3 to 60.1]
Statistical Analysis 1: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q4W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 33.2, 95% CI 2-sided [20.6 to 45.8]
Statistical Analysis 2: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q2W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 37.6, 95% CI 2-sided [26.2 to 49.0]

3. Secondary Outcome: Percent Change in Eczema Area Severity Index (EASI) Score From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  Least Square (LS) Mean was calculated using ANCOVA model with treatment, stratification factors of geographic region, age group, baseline IGA score (IGA 3 versus 4) as fixed factors baseline value as covariate.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 82 | 81 | 123
Percent change | -25.25 (4.765) | -59.74 (4.920) | -64.23 (4.402)
Statistical Analysis 1: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q4W; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -34.50, 95% CI 2-sided [-44.1 to -24.9]
Statistical Analysis 2: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q2W; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -38.99, 95% CI 2-sided [-47.7 to -30.3]

4. Secondary Outcome: Percentage of Participants Achieving EASI-90 at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI-90 responder is defined as a participant who achieves a ≥ 90% reduction from baseline in the EASI score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Induction - Lebrikizumab 250 mg Q4W: Induction Period (Baseline - Week 16): Participants received 500 mg of Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and followed by 250 mg of Lebrikizumab administered SC Q4W from Week 4 until Week 12.
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 82 | 81 | 123
Percentage of participants | 9.8 [3.3 to 16.2] | 28.4 [18.6 to 38.3] | 34.3 [25.9 to 42.7]
Statistical Analysis 1: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q4W; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.4, 95% CI 2-sided [6.8 to 29.9]
Statistical Analysis 2: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q2W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.2, 95% CI 2-sided [13.9 to 34.5]

5. Secondary Outcome: Percentage of Participants With an Itch Numeric Rating Scale (NRS) Score of ≥4-points at Baseline Who Achieve A ≥4-point Reduction From Baseline to Week 1
Description: The Itch Numeric Rating Scale (NRS) is a an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Time Frame: Baseline to Week 1
Population: All randomized participants, with a Baseline Itch NRS Score ≥4, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 60 | 59 | 80
Percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 1.3 [0.0 to 3.7]
Statistical Analysis 1: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q2W; Test type: Superiority; p = 0.404, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.2, 95% CI 2-sided [-1.2 to 3.6]

6. Secondary Outcome: Percentage of Participants With an Itch NRS Score of ≥4-points at Baseline Who Achieve A ≥4-point Reduction From Baseline to Week 2
Description: as for outcome 5
Time Frame: Baseline to Week 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 60 | 59 | 80
Percentage of participants | 0 [0.0 to 0.0] | 1.7 [0.0 to 5.0] | 3.8 [0.0 to 7.9]
Statistical Analysis 1: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q4W; Test type: Superiority; p = 0.294, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.8, 95% CI 2-sided [-1.6 to 5.1]
Statistical Analysis 2: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q2W; Test type: Superiority; p = 0.138, Cochran-Mantel-Haenszel; Risk Difference (RD) = 3.7, 95% CI 2-sided [-0.5 to 7.8]

7. Secondary Outcome: Percentage of Participants With an Itch NRS Score of ≥4-points at Baseline Who Achieve A ≥4-point Reduction From Baseline to Week 4
Description: as for outcome 5
Time Frame: Baseline to Week 4
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 60 | 59 | 80
Percentage of participants | 0 [0.0 to 0.0] | 8.5 [1.4 to 15.6] | 16.3 [8.2 to 24.3]
Statistical Analysis 1: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q4W; Test type: Superiority; p = 0.013, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.2, 95% CI 2-sided [1.8 to 16.5]
Statistical Analysis 2: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q2W; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.2, 95% CI 2-sided [8.1 to 24.3]

8. Secondary Outcome: Percentage of Participants With an Itch NRS Score of ≥4-points at Baseline Who Achieve A ≥4-point Reduction From Baseline to Week 16
Description: as for outcome 5
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250 mg Q4W | Induction - Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 60 | 59 | 80
Percentage of participants | 3.3 [0.0 to 7.9] | 23.8 [12.9 to 34.7] | 32.7 [22.4 to 43.0]
Statistical Analysis 1: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q4W; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.6, 95% CI 2-sided [8.7 to 32.4]
Statistical Analysis 2: Comparison: Induction - Placebo vs Induction - Lebrikizumab 250 mg Q2W; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.2, 95% CI 2-sided [17.9 to 40.4]

ADVERSE EVENTS:
Time Frame: Baseline Up To Week 68.
Description: All randomized participants. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Induction - Lebrikizumab 250mg Q4W: Induction Period (Baseline - Week 16): Participants received 500 mg of Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and followed by 250 mg of Lebrikizumab administered SC Q4W from Week 4 until Week 12.
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250mg Q4W | Induction - Lebrikizumab 250mg Q2W | Maintenance Blinded Period - Lebrikizumab Q4W Responder/Lebrikizumab Q4W | Maintenance Blinded Period - Lebrikizumab Q2W Responder/ Lebrikizumab Q4W | Maintenance Blinded Period - Lebrikizumab Q2W Responder/Lebrikizumab Q2W | Maintenance Blinded Period - Placebo Responder/Placebo | Escape Arm Week 16 - Maintenance Open Label - Placebo Non Responder/Lebrikizumab 250 mg Q2W | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q4W Nonresponder/Lebrikizumab 250mg Q2W | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q2W Nonresponder/Lebrikizumab 250mg Q2W | Escape Arm Week 20 to 64 Maintenance Open Label Lebrikizumab 250 Q2W
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/81 | 0/123 | 0/38 | 0/33 | 0/32 | 0/11 | 0/71 | 0/42 | 0/55 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/82 | 0/81 | 1/123 | 1/38 | 0/33 | 1/32 | 0/11 | 1/71 | 2/42 | 1/55 | 1/8
Other Adverse Events (participants affected / at risk) | 52/82 | 49/81 | 93/123 | 31/38 | 25/33 | 29/32 | 10/11 | 63/71 | 36/42 | 49/55 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction - Placebo (N=82) | Induction - Lebrikizumab 250mg Q4W (N=81) | Induction - Lebrikizumab 250mg Q2W (N=123) | Maintenance Blinded Period - Lebrikizumab Q4W Responder/Lebrikizumab Q4W (N=38) | Maintenance Blinded Period - Lebrikizumab Q2W Responder/ Lebrikizumab Q4W (N=33) | Maintenance Blinded Period - Lebrikizumab Q2W Responder/Lebrikizumab Q2W (N=32) | Maintenance Blinded Period - Placebo Responder/Placebo (N=11) | Escape Arm Week 16 - Maintenance Open Label - Placebo Non Responder/Lebrikizumab 250 mg Q2W (N=71) | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q4W Nonresponder/Lebrikizumab 250mg Q2W (N=42) | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q2W Nonresponder/Lebrikizumab 250mg Q2W (N=55) | Escape Arm Week 20 to 64 Maintenance Open Label Lebrikizumab 250 Q2W (N=8)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/24 (0) | 0/25 (0) | 0/41 (0) | 0/15 (0) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 0/19 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction - Placebo (N=82) | Induction - Lebrikizumab 250mg Q4W (N=81) | Induction - Lebrikizumab 250mg Q2W (N=123) | Maintenance Blinded Period - Lebrikizumab Q4W Responder/Lebrikizumab Q4W (N=38) | Maintenance Blinded Period - Lebrikizumab Q2W Responder/ Lebrikizumab Q4W (N=33) | Maintenance Blinded Period - Lebrikizumab Q2W Responder/Lebrikizumab Q2W (N=32) | Maintenance Blinded Period - Placebo Responder/Placebo (N=11) | Escape Arm Week 16 - Maintenance Open Label - Placebo Non Responder/Lebrikizumab 250 mg Q2W (N=71) | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q4W Nonresponder/Lebrikizumab 250mg Q2W (N=42) | Escape Arm Week 16 Maintenance Open Label-Lebrikizumab 250mg Q2W Nonresponder/Lebrikizumab 250mg Q2W (N=55) | Escape Arm Week 20 to 64 Maintenance Open Label Lebrikizumab 250 Q2W (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blepharitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central serous chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 4 (4) | 10 (11) | 21 (23) | 5 (6) | 1 (1) | 4 (4) | 0 (0) | 13 (14) | 1 (1) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Eye opacity (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye paraesthesia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Giant papillary conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pingueculitis (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 5 (5) | 2 (3) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2) | 1 (2) | 2 (7) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (3) | 3 (34) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site paraesthesia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 1 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 3 (11) | 0 (0) | 2 (14) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (29) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 13 (15) | 15 (18) | 25 (32) | 7 (11) | 6 (6) | 11 (15) | 3 (3) | 13 (14) | 4 (5) | 5 (5) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 4 (4) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholinitis (Infections and infestations) | 0/24 (0) | 0/25 (0) | 0/41 (0) | 1/15 (1) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 0/19 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 5 (5) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 10 (13) | 1 (2) | 1 (1) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 7 (7) | 7 (8) | 4 (4) | 0 (0) | 13 (13) | 8 (8) | 12 (13) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (8) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 8 (8) | 5 (5) | 7 (7) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 2 (6) | 5 (6) | 1 (2)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 2 (2) | 1 (1) | 1 (2) | 3 (6) | 3 (10) | 1 (1) | 0 (0) | 2 (3) | 8 (11) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malassezia infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5) | 7 (8) | 2 (4) | 2 (3) | 3 (3) | 1 (1) | 8 (8) | 6 (7) | 7 (8) | 1 (1)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (3) | 2 (2) | 6 (6) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 0 (0)
Otitis externa (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urogenital infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1/24 (1) | 0/25 (0) | 0/41 (0) | 0/15 (0) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 0/19 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluoride increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hormone level abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 8 (8) | 2 (2) | 4 (4) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 5 (8) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 3 (4) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (2) | 1 (1) | 2 (2) | 3 (5) | 4 (4) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslalia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (16) | 3 (4) | 4 (7) | 1 (1) | 6 (16) | 4 (4) | 1 (1) | 4 (17) | 2 (3) | 2 (4) | 1 (5)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstrual headache (Nervous system disorders) | 1/24 (2) | 0/25 (0) | 0/41 (0) | 0/15 (0) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 1/19 (1) | 0/9 (0) | 0/15 (0) | 0/3 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0/24 (0) | 0/25 (0) | 0/41 (0) | 0/15 (0) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 0/19 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/24 (0) | 0/25 (0) | 2/41 (2) | 0/15 (0) | 2/12 (2) | 1/12 (1) | 0/5 (0) | 2/19 (7) | 0/9 (0) | 1/15 (1) | 0/3 (0)
Endometriosis (Reproductive system and breast disorders) | 0/24 (0) | 1/25 (1) | 0/41 (0) | 0/15 (0) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 0/19 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1/24 (1) | 0/25 (0) | 0/41 (0) | 0/15 (0) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 0/19 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/24 (0) | 0/25 (0) | 0/41 (0) | 0/15 (0) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 0/19 (0) | 0/9 (0) | 1/15 (1) | 0/3 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 4 (4) | 1 (1) | 6 (6) | 3 (3) | 1 (1) | 5 (6) | 3 (3) | 6 (8) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chloasma (Skin and subcutaneous tissue disorders) | 0/24 (0) | 1/25 (1) | 0/41 (0) | 0/15 (0) | 0/12 (0) | 0/12 (0) | 0/5 (0) | 0/19 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Needle track marks (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Anal fistula repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental care (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 1 (1)
Tooth restoration (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT04760314/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT04760314/SAP_001.pdf